CLINICAL TRIAL: NCT00868608
Title: A Phase 2 Study Of Inotuzumab Ozogamicin (Cmc-544) In Subjects With Indolent Non-hodgkin's Lymphoma (Nhl) That Is Refractory To Or Has Relapsed After Rituximab And Chemotherapy Or Radioimmunotherapy
Brief Title: Study Evaluating Inotuzumab Ozogamicin (CMC-544) In Indolent Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 3129K7-2001; B1931007 (Other: Alias Study Number); 2008-001635-34 (EudraCT Number)
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma
Keywords: Refractory Indolent NHL; lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- inotuzumab ozogamicin (Experimental): inotuzumab ozogamicin
  Interventions: Drug: Inotuzumab Ozogamicin (CMC-544)

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin (CMC-544) — Administered intravenously at 1.8 mg/m2 every 4 weeks for a planned 4 - 8 cycles
  Other Names: inotuzumab ozogamicin

SUMMARY:
The purpose of this study is to evaluate the efficacy of inotuzumab ozogamicin (CMC-544) in subjects with indolent Non-Hodgkins lymphoma (NHL) that is refractory or has relapsed after multiple therapies including rituximab or radioimmunotherapy. The investigational drug will be given to subjects with indolent NHL by intravenous infusion at a dose of 1.8 mg/m2, every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been previously diagnosed with CD22-positive, indolent NHL (defined as follicular, marginal zone, or small lymphocytic lymphoma) that has progressed after 2 or more prior systemic therapies.
* Previous anticancer treatment given must have contained rituximab and chemotherapy, or anti CD20 Radio Immuno Therapy. Subjects must have exhibited no response or have progressed within 6 months from the completion of the most recent rituximab or rituximab containing therapy or within 12 months of the completion of Radio Immuno Therapy.
* Measurable disease with adequate bone marrow function, renal and hepatic function

Exclusion Criteria:

* History of, or suggestive of, veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS) or history of chronic liver disease (eg, cirrhosis) or suspected alcohol abuse.
* Prior allogeneic hematopoietic stem cell transplant (HSCT).
* Clinical evidence of transformation to a more aggressive subtype of lymphoma or grade 3b follicular lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-07-30 (Actual); Primary Completion 2012-01-10 (Actual); Study Completion 2013-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (22):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Loma Linda University Cancer Center, Loma Linda, California
  - Loma Linda University Cancer Center #5, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Facey Medical Group, Mission Hills, California
  - Providence Holy Cross, Mission Hills, California
  - Rush University Medical Center, Chicago, Illinois
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - New York Medical College, Hawthorne, New York
  - Quest Diagnostics, Allentown, Pennsylvania
  - Carlisle Regional Medical Center Lab, Carlisle, Pennsylvania
  - Penn State Milton S. Hershey medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CMSA Medical Lab, State College, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen UZ Gasthuisberg, Leuven
  - Oncologisch Centrum GZA - Location St. Augustinus, Wilrijk
- Germany (2):
  - Charite Campus Mitte, Berlin
  - Charite Berlin-Campus Virchow-Klinikum, Berlin
- The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, N.T., Hong Kong
- Hungary (2):
  - Debreceni Egyetem Orvos-es Egeszsegtudomanyi Centrum Belgyogyaszati Intezet,, Debrecen
  - Kaposi Mor Oktato Korhaz, Belgyogyaszati Osztaly, Kaposvár
- Japan (8):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - EPMint Co., Ltd, Aichi
  - Nagoya Daini Red Cross Hospital, Aichi
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hp. Org. Kyushu Medical Center, Fukuoka
  - Tokai University Hospital, Kanagawa
  - Cancer Inst. Hp. of Japanese Foundation for Cancer Research, Tokyo
- Netherlands (2):
  - Erasmus Medisch Centrum, Rotterdam
  - Erasmus MC Apotheek, Rotterdam
- Singapore General Hospital, Singapore, Singapore
- Samsung Medical Center, Seoul, Korea, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K7-2001&StudyName=Study%20Evaluating%20Inotuzumab%20Ozogamicin%20%28CMC-544%29%20In%20Indolent%20Non-Hodgkins%20Lymphoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Inotuzumab Ozogamicin - NHL Type (Follicular): Participants who have been previously diagnosed with CD22-positive, indolent Non-Hodgkin's Lymphoma (NHL) defined as follicular (the most common of the indolent B-cell lymphomas, comprising approximately 22 percent [%] of all B-cell lymphomas) received inotozumab ozogamicin, administered at 1.8 milligrams per square meter (mg/m^2) intravenously (IV) on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles. After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
- Inotuzumab Ozogamicin - NHL Type (Marginal Zone): Participants who have been previously diagnosed with CD22-positive, indolent NHL defined as marginal zone (a less common form of indolent B-cell lymphomas, comprising approximately 6% of all B-cell lymphomas) received inotozumab ozogamicin, administered at 1.8 mg/m^2 IV on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles. After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
- Inotuzumab Ozogamicin - NHL Type (Small Lymphocytic): Participants who have been previously diagnosed with CD22-positive, indolent NHL defined as small lymphocytic (a less common form of indolent B-cell lymphomas, comprising approximately 5% of all B-cell lymphomas) received inotozumab ozogamicin, administered at 1.8 mg/m^2 IV on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles. After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular) | Inotuzumab Ozogamicin - NHL Type (Marginal Zone) | Inotuzumab Ozogamicin - NHL Type (Small Lymphocytic)
Started | 72 | 4 | 5
Completed | 49 | 1 | 0
Not Completed | 23 | 3 | 5
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Lost to Follow-up | 3 | 0 | 1
Not completed — Death | 16 | 2 | 4
Not completed — Other - Unspecified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inotuzumab Ozogamicin - NHL Type (Follicular): Participants who have been previously diagnosed with CD22-positive, indolent NHL defined as follicular (the most common of the indolent B-cell lymphomas, comprising approximately 22 % of all B-cell lymphomas) received inotozumab ozogamicin, administered at 1.8 mg/m^2 IV on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles. After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular) | Inotuzumab Ozogamicin - NHL Type (Marginal Zone) | Inotuzumab Ozogamicin - NHL Type (Small Lymphocytic) | Total
Number analyzed (Participants) | 72 | 4 | 5 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (10.2) | 70.8 (13.5) | 65.2 (10.0) | 61.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 2 | 0 | 37
  Male | 37 | 2 | 5 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Indolent NHL Achieving CR or Partial Response (PR) According to International Response Criteria for NHL
Description: CR was defined as complete disappearance of all target lesions and disease-related symptoms; all nodes must have decreased to normal (less than or equal to [≤]1.5 cm in their greatest transverse diameter [GTD] for nodes more than [>]1.5 cm before therapy) or ≤1 cm (short axis) in previously involved node; enlarged spleen prior to therapy must have regressed and be non-palpable; bone marrow lymphoma: infiltrate must have been cleared on repeat bone marrow aspirate and biopsy. PR was defined as >50% decrease in the sum of the product diameters (SPD) of up to 6 index lesions. No increase in size of other nodes, liver or spleen. Splenic and hepatic nodules must have regressed by greater than or equal to [≥]50% in the SPD or GTD (for single nodules). With exception of splenic and hepatic nodules, involvement of other organs was usually assessable and no measurable disease should be present. No progression of non-target disease or new lesions.
Time Frame: Assessed for up to 2 years, including planned assessments every 8 to 12 weeks from first dose of study drug. Follow-up period may have been extended beyond 2 years due to dosing delays and allowed study visit windows.
Population: Intent to treat (ITT) population: all participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Inotuzumab Ozogamicin - Total (All NHL Types): Participants who have been previously diagnosed with CD22-positive, indolent NHL (defined as follicular, marginal zone or small lymphocytic lymphoma) received inotozumab ozogamicin, administered at 1.8 mg/m^2 IV on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles. After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Percentage of Participants | 66.7 [55.32 to 76.76]

2. Secondary Outcome: Percentage of Participants With Follicular NHL Achieving CR or PR According to International Response Criteria for NHL
Description: CR was defined as complete disappearance of all target lesions and disease-related symptoms; all nodes must have decreased to normal (≤1.5 cm in their greatest transverse diameter for nodes >1.5 cm before therapy) or ≤1 cm (short axis) in previously involved node; enlarged spleen prior to therapy must have regressed and be non-palpable; bone marrow lymphoma: infiltrate must have been cleared on repeat bone marrow aspirate and biopsy. PR was defined as >50% decrease in the SPD of up to 6 index lesions. No increase in size of other nodes, liver or spleen. Splenic and hepatic nodules must have regressed by ≥50% in the SPD or greatest transverse diameter (for single nodules). With exception of splenic and hepatic nodules, involvement of other organs was usually assessable and no measurable disease should be present. No progression of non-target disease or new lesions.
Time Frame: as for outcome 1
Population: ITT population (participants with NHL type defined as follicular).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Inotuzumab Ozogamicin - NHL Type (Follicular): Participants who have been previously diagnosed with CD22-positive, indolent NHL defined as follicular (the most common of the indolent B-cell lymphomas, comprising approximately 22% of all B-cell lymphomas) received inotozumab ozogamicin, administered at 1.8 mg/m^2 IV on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles. After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 72
Percentage of Participants | 70.8 [58.93 to 80.95]

3. Secondary Outcome: Percentage of Participants With Indolent NHL Achieving a CR According to International Response Criteria for NHL
Description: CR was defined as complete disappearance of all target lesions and disease-related symptoms; all nodes must have decreased to normal (≤1.5 cm in their greatest transverse diameter for nodes >1.5 cm before therapy) or ≤1 cm (short axis) in previously involved node; enlarged spleen prior to therapy must have regressed and be non-palpable; bone marrow lymphoma: infiltrate must have been cleared on repeat bone marrow aspirate and biopsy.
Time Frame: as for outcome 1
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Percentage of Participants | 30.9 [21.07 to 42.11]

4. Secondary Outcome: Percentage of Participants With Follicular NHL Achieving a CR According to International Response Criteria for NHL
Description: as for outcome 3
Time Frame: as for outcome 1
Population: ITT population (participants with NHL type defined as follicular).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Inotuzumab Ozogamicin - NHL Type (Follicular): Participants who have been previously diagnosed with CD22-positive, indolent NHL defined as follicular (the most common of the indolent B-cell lymphomas, comprising approximately 22% of all B-cell lymphomas) received inotozumab ozogamicin, administered at 1.8 mg/m^2 IV on Day 1 of each 28-day cycle for at least 4 cycles and up to a maximum of 8 cycles (in participants who achieved a CR). After Cycle 1, the dose and/or the frequency may have been adjusted, based on toxicities. Participants who may have derived benefit from additional treatment may have continued to receive additional cycles of test article, up to a maximum of 2 additional cycles after achievement of a CR or up to a maximum of 8 cycles, whichever occurred first.
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 72
Percentage of Participants | 34.7 [23.88 to 46.86]

5. Secondary Outcome: Duration of Response in Participants With Indolent NHL
Description: Duration of response was measured from the first date of response until the first date that the objective progression of disease (PD) or symptomatic deterioration or initiation of new anticancer therapy for the lymphoma or death from any cause is documented. Participants without an event were censored at the date of the last valid tumor assessment. A valid tumor assessment visit was defined as the tumor assessment visit with overall response of CR, PR, stable disease (SD), or PD, but not 'Not Done' or 'Unknown'. PD was defined according to the International Response Criteria for NHL: 1) New lesion or increase by ≥50% of previously involved sites from nadir, 2) New lesion(s) >1.5 cm (any axis); ≥50% increase in SPD of >1 node; or ≥50% increase in longest diameter of previously identified node >1 cm in short axis, 3) >50% increase from nadir in the SPD of any previous lesions (splenic or hepatic) and 4) New or recurrent involvement in bone marrow.
Time Frame: as for outcome 1
Population: Participants with Indolent NHL who responded.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 54
Months | 24.8 [10.9 to NA] — Upper confidence interval (CI) could not be estimated by the SAS LIFETEST procedure due to limited number of events observed. SAS LIFETEST is a statistical procedure used to make inferences about a broader population based on the sample data.

6. Secondary Outcome: Probability of Maintaining a Response at 6, 12 and 24 Months in Participants With Indolent NHL
Description: Duration of response was measured from the first date of response until the first date that the objective PD or symptomatic deterioration or initiation of new anticancer therapy for the lymphoma or death from any cause is documented. Participants without an event were censored at the date of the last valid tumor assessment. A valid tumor assessment visit was defined as the tumor assessment visit with overall response of CR, PR, stable disease (SD), or PD, but not 'Not Done' or 'Unknown'. PD was defined according to the International Response Criteria for NHL: 1) New lesion or increase by ≥50% of previously involved sites from nadir, 2) New lesion(s) >1.5 cm (any axis); ≥50% increase in SPD of >1 node; or ≥50% increase in longest diameter of previously identified node >1 cm in short axis, 3) >50% increase from nadir in the SPD of any previous lesions (splenic or hepatic) and 4) New or recurrent involvement in bone marrow.
Time Frame: 6, 12 and 24 months
Population: Participants with Indolent NHL who responded.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 54
Probability
  6 Month Probability of Maintaining a Response | 0.82 [0.68 to 0.90]
  12 Month Probability of Maintaining a Response | 0.65 [0.50 to 0.77]
  24 Month Probability of Maintaining a Response | 0.53 [0.38 to 0.66]

7. Secondary Outcome: Duration of Response in Participants With Follicular NHL
Description: as for outcome 6
Time Frame: as for outcome 1
Population: Participants with Follicular NHL who responded.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 51
Months | 24.8 [12.9 to NA] — Upper CI could not be estimated by the SAS LIFETEST procedure due to limited number of events observed. SAS LIFETEST is a statistical procedure used to make inferences about a broader population based on the sample data.

8. Secondary Outcome: Probability of Maintaining a Response at 6, 12 and 24 Months in Participants With Follicular NHL
Description: as for outcome 6
Time Frame: 6, 12 and 24 months
Population: Participants with Follicular NHL who responded.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 51
Probability
  6 Month Probability of Maintaining a Response | 0.85 [0.71 to 0.92]
  12 Month Probability of Maintaining a Response | 0.67 [0.51 to 0.79]
  24 Month Probability of Maintaining a Response | 0.57 [0.40 to 0.70]

9. Secondary Outcome: Kaplan-Meier Estimate of the Progression-Free Survival (PFS) in Participants With Indolent NHL
Description: Kaplan-Meier: a rule for calculating an estimate of survival. PFS was defined as time from enrollment to death from any cause without progression, progression during and after treatment, and initiation of all new anti-cancer treatments for the lymphoma. For participants with no event, censorship occurred at the date of last valid disease assessment. PD was defined in accordance with the International Response Criteria for NHL: 1) New lesion or increase by ≥50% of previously involved sites from nadir, 2) New lesion(s) >1.5 cm (any axis); ≥50% increase in SPD of >1 node; or ≥50% increase in longest diameter of previously identified node >1 cm in short axis, 3) >50% increase from nadir in the SPD of any previous lesions (splenic or hepatic) and 4) New or recurrent involvement in bone marrow.
Time Frame: as for outcome 1
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Months | 12.7 [8.9 to 26.9]

10. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Alive and Free From PD or New Anticancer Therapy at 6, 12 and 24 Months in Participants With Indolent NHL
Description: as for outcome 9
Time Frame: 6, 12 and 24 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Percent Probability
  6 Months | 65.1 [53.3 to 74.6]
  12 Months | 52.0 [40.0 to 62.7]
  24 Months | 41.3 [29.8 to 52.5]

11. Secondary Outcome: Kaplan-Meier Estimate of the PFS in Participants With Follicular NHL
Description: Kaplan-Meier: a rule for calculating an estimate of survival. PFS was defined as time from enrollment to progression of disease or death from any cause. Events were defined as death from any cause without progression, progression during and after treatment, and initiation of all new anti-cancer treatments for the lymphoma. For participants with no event, censorship occurred at the date of last valid disease assessment. PD was defined in accordance with the International Response Criteria for NHL: 1) New lesion or increase by ≥50% of previously involved sites from nadir, 2) New lesion(s) >1.5 cm (any axis); ≥50% increase in SPD of >1 node; or ≥50% increase in longest diameter of previously identified node >1 cm in short axis, 3) >50% increase from nadir in the SPD of any previous lesions (splenic or hepatic) and 4) New or recurrent involvement in bone marrow.
Time Frame: as for outcome 1
Population: ITT population (participants with NHL type defined as follicular).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 72
Months | 14.7 [11.0 to NA] — Upper CI could not be estimated by the SAS LIFETEST procedure due to limited number of events observed. SAS LIFETEST is a statistical procedure used to make inferences about a broader population based on the sample data.

12. Secondary Outcome: Kaplan-Meier Estimate of the Probability of Being Alive and Free From PD or New Anticancer Therapy at 6, 12 and 24 Months in Participants With Follicular NHL
Description: as for outcome 11
Time Frame: 6, 12 and 24 months
Population: ITT population (participants with NHL type defined as follicular).
Measure: Number (95% Confidence Interval); unit: Percenr probability
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 72
Percenr probability
  6 Months | 69.3 [56.8 to 78.8]
  12 Months | 56.3 [43.4 to 67.3]
  24 Months | 46.1 [33.5 to 57.8]

13. Secondary Outcome: Kaplan-Meier Estimate of the Overall Survival (OS) in Participants With Indolent NHL
Description: Kaplan-Meier: a rule for calculating an estimate of survival. OS was defined as the time from enrollment to death from any cause. For participants without death, censorship occurred at the date of last contact.
Time Frame: Any time up to 2 years after enrollment. Follow-up period may have been extended beyond 2 years due to dosing delays and allowed study visit windows.
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Months | NA [26.6 to NA] — Median and upper CI could not be estimated by the SAS LIFETEST procedure due to limited number of events observed. SAS LIFETEST is a statistical procedure used to make inferences about a broader population based on the sample data.

14. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Survival at 6, 12 and 24 Months in Participants With Indolent NHL
Description: as for outcome 13
Time Frame: 6, 12 and 24 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Probability
  6 Months | 0.89 [0.79 to 0.94]
  12 Months | 0.80 [0.69 to 0.87]
  24 Months | 0.73 [0.61 to 0.81]

15. Secondary Outcome: Kaplan-Meier Estimate of the OS in Participants With Follicular NHL
Description: as for outcome 13
Time Frame: as for outcome 13
Population: ITT population (participants with NHL type defined as follicular).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 72
Months | NA [NA to NA] — Median and lower and upper CIs could not be estimated by the SAS LIFETEST procedure due to limited number of events observed. SAS LIFETEST is a statistical procedure used to make inferences about a broader population based on the sample data.

16. Secondary Outcome: Kaplan-Meier Esitmates of the Probability of Survival at 6, 12 and 24 Months in Participants With Follicular NHL
Description: as for outcome 13
Time Frame: 6, 12 and 24 months
Population: ITT population (participants with NHL type defined as follicular).
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular)
Number analyzed (Participants) | 72
Probability
  6 Months | 0.91 [0.82 to 0.96]
  12 Months | 0.83 [0.72 to 0.90]
  24 Months | 0.78 [0.67 to 0.86]

17. Secondary Outcome: Median Induced Change From Baseline of QT Study Specific Correction (QTcS) by Cycle Based on Median Maximum Calicheamicin Concentration (Cmax)
Description: Triplicate 12-lead electrocardiogram (ECG) measurements were performed approximately 2 minutes apart. ECG assessments were pre-specified in the protocol to be time-matched with selected pharmacokinetic (PK) samples in order to conduct a concentration-QTc analysis. A study-specific QT correction factor was estimated using the un-averaged triplicate data and was used to calculate the study-specific corrected QT (QTcS). QTcS interval versus serum concentrations were modeled using a population analysis approach to identify potential effects of total calicheamicin exposure. Results for drug effects were based on the median Cmax for total calicheamicin across all participants: median Cmax was 61.3 ng/mL
Time Frame: Cycle 1: pre-dose, 1 hour; Cycle 3 & 4: pre-dose, 1, 3, 48, 168 hours; Cycle 6 (if applicable): pre-dose; end of treatment: during clinic visit
Population: There were 80 participants in the analysis dataset, but time-matched PK-ECG data only existed for 73 participants (35 female).
Measure: Median (90% Confidence Interval); unit: Milliseconds (msec)
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 80
Milliseconds (msec)
  Cycle 1 | 3.51 [1.85 to 5.40]
  Cycle 2 | 5.00 [3.19 to 6.80]
  Cycle 3 | 6.41 [4.01 to 8.64]
  Cycle 4 | 7.83 [4.83 to 10.8]

18. Secondary Outcome: Percentage of Participants With a Treatment Emergent Adverse Event (TEAE) (Safety Population)
Description: Includes all TEAEs: any event that emerged after the first dose of the study treatment during the treatment period that was absent before administration of any study treatment, or worsened during the treatment period relative to the pre-treatment state.
Time Frame: Protocol reporting period: from informed consent to at least 28 days after the last dose.
Population: Safety Population - includes all participants who received at least 1 dose of study medication. This population only excluded participants who never received any study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Percentage of Participants
  % participants with a TEAE | 96.3
  % participants with serious TEAE | 18.5
  % participants with Grade 3 or higher TEAE | 77.8
  % participants for study drug discontinuation | 58.0
  % participants with dose reduction due to TEAE | 33.3
  % participants for study drug stopped temporarily | 48.1

19. Secondary Outcome: Percentage of Participants With QTc Interval Corrected Using Fridericia's Formula (QTcF) by Category (Safety Population)
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to the beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR). Maximum QTcF was categorized as less than or equal to (≤) 450 msec, >450 msec to ≤480 msec, >480 msec to ≤500 msec and >500 msec. Participants are reported only once under the maximum QTcF interval observed at any of the time-points. Maximum increase from baseline was categorized as <30 msec, ≥30 to <60 msec (borderline) and ≥60 msec (prolonged) were summarized.
Time Frame: Screening; Cycle 1: pre-dose & 1 hour; Cycles 3 and 4: pre-dose, 1, 3, 48, and 168 hours; Cycle 6: pre-dose; end of treatment: 28 to 56 days post-last dose.
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin - Total (All NHL Types)
Number analyzed (Participants) | 81
Percentage of Participants
  % participants with QTcF ≤450 ([msec) | 83.1
  % participants with QTcF >450 to ≤480 (msec) | 14.3
  % participants with QTcF >480 to ≤500 (msec) | 2.6
  % participants with QTcF >500 (msec) | 0
  % participants with any baseline increase | 98.7
  % participants baseline increase <30 (msec) | 79.2
  % participants baseline increase ≥30 to <60 (msec) | 18.2
  % participants baseline increase ≥60 (msec) | 1.3

ADVERSE EVENTS:
Time Frame: Collected from time of informed consent up to a minimum of 28 days after last dose of study drug. Adverse event (AE) summaries below are inclusive of AEs from first dose.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Inotuzumab Ozogamicin - NHL Type (Follicular) | Inotuzumab Ozogamicin - NHL Type (Marginal Zone) | Inotuzumab Ozogamicin - NHL Type (Small Lymphocytic)
Serious Adverse Events (participants affected / at risk) | 12/72 | 2/4 | 1/5
Other Adverse Events (participants affected / at risk) | 69/72 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin - NHL Type (Follicular) (N=72) | Inotuzumab Ozogamicin - NHL Type (Marginal Zone) (N=4) | Inotuzumab Ozogamicin - NHL Type (Small Lymphocytic) (N=5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Sepsis (Infections and infestations) | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Budd-Chiari syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin - NHL Type (Follicular) (N=72) | Inotuzumab Ozogamicin - NHL Type (Marginal Zone) (N=4) | Inotuzumab Ozogamicin - NHL Type (Small Lymphocytic) (N=5)
Anaemia (Blood and lymphatic system disorders) | 12 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 26 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 25 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 40 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 55 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 35 | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 14 | 0 | 1
Chills (General disorders) | 6 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 34 | 3 | 2
Oedema peripheral (General disorders) | 7 | 0 | 0
Pyrexia (General disorders) | 14 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 5 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 16 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 32 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 21 | 1 | 0
Blood chloride increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 5 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 5 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 21 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Monocyte count increased (Investigations) | 2 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 4 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 11 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 20 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 0 | 1
Dysgeusia (Nervous system disorders) | 5 | 0 | 0
Headache (Nervous system disorders) | 12 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 0 | 0

LIMITATIONS AND CAVEATS:
The sample size for this study was determined by clinical rather than statistical considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less